CLINICAL TRIAL: NCT06492343
Title: Real Time Neurofeedback, Its Neurotransmitter Underpinnings, and Therapeutic Effects, in Clinical High Risk Individuals
Brief Title: Neurofeedback in Clinical High Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 206731
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Real Neurofeedback From DMN; Sham Neurofeedback From Motor Cortex
Keywords: fMRI, neurofeedback, DMN, functional connectivity

STUDY DESIGN:
Intervention Model Description: one group receiving NFB from DMN another group receiving NFB from motor cortex
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real NFB from DMN (Experimental): Participants will receive NFB from their DMN
  Interventions: Other: fMRI based neurofeedback
- sham NFB from motor cortex (Experimental): Participants will receive NFB from their motor cortex
  Interventions: Other: fMRI based neurofeedback

INTERVENTIONS:
Other: fMRI based neurofeedback — participants will receive neurofeedback from their brain in order to modify their own brain function

SUMMARY:
The goal of this trial is to test whether fMRI based neurofeedback from default mode network (DMN) will reduce DMN hyperconnectivity in clinical high risk individuals, which will lead to reductions in clinical symptoms and improve cognitive performance.

DETAILED DESCRIPTION:
Identification of brain abnormalities in first episode schizophrenia (SZ) patients has provided evidence that disease-related abnormalities develop prior to psychosis and helped shift attention to the identification of a prepsychotic,clinical high risk (CHR) for psychosis prodromal period 11,12 A recent meta-analysis showed that CHR individuals have an elevated risk for developing psychosis of 11% after 6 months, 15% after 12 months, 20% after 24 months, and 23% after 36 months8. Furthermore, our work and others demonstrate that CHR individuals show deficits in both brain function and cognition similar to those in SZ 1,8. These include default mode network (DMN) hyper-connectivity, (between medial prefrontal cortex (MPFC) and posterior cingulate cortex (PCC)) and reduced MPFC-dorsolateral prefrontal cortex (DLPFC: part of a central executive network (CEN)) anticorrelation in CHR, similar to findings reported in SZ. These results not only point to a way in which abnormal brain function contributes to SZ development, but also motivate the search for approaches to alter the disease trajectory. Thus, in the R61 portion of the current application, we will examine the efficacy of mindfulness meditation augmented, real-time-fMRI-neurofeedback (rt-NFB) in reducing DMN hyperconnectivity and increasing MPFC-DLPFC anticorrelations, post-NFB, similar to what we observed in chronic SZ, and assess glutamate (Glu) and gammaaminobutyric acid (GABA) levels in MPFC, PCC, and DLPFC. In the R33, we will test the rt-NFB efficacy in a larger sample, examine the relationship between rt-NFB mediated neural network changes and behavioral measures (reductions in symptoms and improvement in working memory (WM)/attentional function). We will also examine cellular level changes via magnetic resonance spectroscopy (MRS) measures of Glu and GABA to arrive at a more comprehensive understanding of what cellular phenomena underlie rt-NFB. This application builds on three sources of evidence: 1. Fogarty grant (PI: Stone, co-PI: Niznikiewicz, Whitfield-Gabrieli) showing MPFC-PCC hyperconnectivity and its correlations with SIPS scores in CHR (see preliminary data (PD)); 2. R21 results (PI: Niznikiewicz) showing that rt-NFB can reduce BOLD activation in the superior temporal gyrus (STG) 13, and hyperconnectivity in DMN 14 in SZ, which in turn were associated with a reduction in auditory hallucinations (AH); and 3. R61/33 (mPI: Niznikiewicz, Whitfield-Gabrieli) ) that confirmed that rt-NFB can modulate DMN connectivity and STG activation in SZ with AH. Based on our PD and the existing literature, in R61, we propose that: 1) rt-NFB directed at DMN will lead to MPFC-PCC hyper-connectivity reductions and an increase in MPFC-DLPFC anticorrelations. For R33 we propose to 1). confirm these findings in a larger independent sample 2) show that improvements in MPFCPCC hyper-connectivity, and MPFC-DLPFC anticorrelations will lead to improvements in clinical symptoms and cognition respectively; and 3) changes in resting state (rs) connectivity will be related to changes in Glu and GABA levels, post-rt-NFB, as assessed by co-localized cellular and connectivity changes pre- vs post-rt-NFB.

R61 PHASE: Overview: We will demonstrate brain target engagement, i.e., the MPFC-PCC rsconnectivity reduction. We will test 40 CHR randomized to 1) one session of rt- NFB directed at DMN (real-rt-NFB; N=20) 2) sham-rt-NFB (N=20) (rt-NFB derived from the motor cortex activation). We will test 20 HC as a benchmark comparison group. The MFC-PCC rs-connectivity reduction in the real rt-NFB group post-rt-NFB, will be the R61 GO criterion. We will also collect MRS data from the MPFC, PCC, and DLPFC.

Aim 1: Brain target engagement using rt-NFB. Based on PD, we predict DMN rs-connectivity reduction in the real rt-NFB group receiving rt-NFB from the DMN-CEN, but not in the sham rt-NFB group. (R61 GO criteria).

Aim 2: Measure Glu and GABA (exploratory) in MPFC, PCC, and DLPFC voxels of interest (VOI). R33 PHASE: Overview: In CHR, we will use a randomized trial, with partial cross-over design: CHR will be randomized to real rt-NFB (N=30), or one sham rt-NFB (N=30) session, followed by real rt-NFB session.; 30 HCs will be scanned once. MRS in the two VOIs will be recorded before and after each rt-NFB session (either real or sham). We will replicate the R61 findings and relate them to clinical and cognitive data. The R33 GO criteria (for future studies): replicating R61 results, significant clinical symptom reductions related to MPFC-PCC connectivity reduction and cognitive improvement related to MPFC-DLPFC anticorrelations increase, post-rt-NFB.

Aim 1: Replicate the R61 Aim 1: We predict that DMN-directed rt-NFB will result in MPFC-PCC rs-connectivity reduction, and MPFC-DLPFC increased anticorrelation in the real rt-NFB group only.

Aim 2: Demonstrate association between DMN rs-connectivity and clinical changes and MPFC-DLPFC anticorrelations and cognitive changes, post-rtfMRI. We predict: associations between 1) reductions of MPFC-PCC connectivity and reductions of SIPS scores, and 2) MPFC-DLPFC anticorrelations increases and WM/attentional improvements in the real rt-NFB group only (see PD).

Aim 3: Co-localization of MRS and fMRI data: Measure Glu and GABA in two selected, individually defined VOIs (based on rs-data) before and after rt-NFB in CHR and HC at baseline.

Aim 4: (exploratory) Correlate Glu/GABA (see Aim 3 for VOIs definitions) with rs-connectivity and clinical and cognitive data, post-rt-NFB. Based on our PD, we predict 1) positive associations between MPFC GABA levels and MPFC-DLPFC anti-correlations, and WM/attention improvements. 2) Glu/GABA ratios associations with MPFC-PCC connectivity reductions, and SIPS scores reductions.

ELIGIBILITY:
Inclusion Criteria:

* For CHR Inclusion:

  1. 12-30 years old
  2. Native speaker or early learner (by age of 6) of English
  3. COPS diagnostic criteria met For HC Inclusion

  <!-- -->

  1. 12-30 years old
  2. Native speaker or early learner (by age of 6) of English
  3. Provides a match with CHR subject on demographic matching variables

     Exclusion Criteria:

     For CHR:

     Exclusion:

  <!-- -->

  1. Meeting DSM-5 criteria for lifetime psychotic disorder, including affective psychoses
  2. WASI-II IQ < 70
  3. Psychosis risk symptoms caused by other psychiatric disorders (including substance use/misuse)
  4. Congenital or acquired CNS disorder that could account for psychosis-risk or cognitive symptoms
  5. Medication that interferes with assessment / presentation of psychosis risk or that could account for psychosis risk symptoms
  6. Antipsychotic medication administered in the absence of evidence the individual was still in the CHR state when treatment began
  7. Inability or refusal to provide informed consent

     For HC:

  <!-- -->

  1. Meets criteria for a psychosis-risk syndrome
  2. Current or previous diagnosis for psychotic di sorder
  3. DSM-5 Cluster A personality disorder
  4. First degree biological relative with psychotic disorder or psychotic symptoms
  5. Current use of psychotropic medication
  6. WASI-II IQ <70
  7. Congenital or acquired CNS disorder that interferes with cognition or produces psychosis risk-like symptoms
  8. Inability or refusal to provide informed consent

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
rs-FMRI DMN changes, post-NFB | three weeks
  reductions in resting state functional connectivity MPFC-PPC in real NFB group only
rs fMRI MPFC-STG changes, post-NFB | three weeks
  reductions in MPFC-PCC resting state functional connectivity, post NFB, in real NFB group only

SECONDARY OUTCOMES:
GABA in MPFC | one week
  GABA levels at baseline in MPFC

CONTACTS AND LOCATIONS:
Overall Officials: margaret niznikiewicz, phd, Principal Investigator — Boston VA Research Institute, Inc.